CLINICAL TRIAL: NCT00426231
Title: Culturally-Tailored Hospital-based Model to Improve Statin Use and Outcomes in Patients With Coronary Disease
Brief Title: Culturally-Tailored Approach to Improve Medication Use in Patients With Heart Attacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Dhananjay Vaidya, Associate Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NA_00001948; AHA 0670015N
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Arteriosclerosis; Myocardial Infarction
Keywords: Randomized Controlled Trials; Health Education; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Patient Nonadherence
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Health Education; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Navigator intervention (Experimental): Patient Navigator intervention
  Interventions: Behavioral: Navigation by a health worker
- Information control (Active Comparator): Information control
  Interventions: Behavioral: Information control

INTERVENTIONS:
Behavioral: Navigation by a health worker — Help provided by health worker to navigate medication access programs
  Arms: Patient Navigator intervention
Behavioral: Information control — Information about medication access programs provided to the participant and their healthcare provider
  Other Names: Enhanced usual care
  Arms: Information control

SUMMARY:
Our research aims to improve the use of medicines known to prevent recurrent heart attacks. In particular, we know that statin treatment is useful after heart attacks, but many patients do not use it. There are a few possible reasons for this. Patients cannot find affordable medicine. Their doctor may not prescribe the medicine after they leave the hospital. Some people may culturally mistrust using the medicine. So they may decide not to take it even if it is prescribed. We are developing a hospital based culturally attuned program to target this problem. In this program, a community health worker counsels and helps patients in accessing pharmacy assistance programs. We will test whether this program can improve appropriate statin use.

We will enroll patients who have heart attacks. We will compare patients who are counseled by the community health worker with those who get the usual care at baseline and at 6 and 12 months (participants enrolled during the early phase of the recruitment will have an additional study visit at 24 months). We will test if their "bad" cholesterol levels are controlled. We will find out how regularly they have filled their questionnaire and taken the medicine. Finally, we will test if they are getting benefit from the statin treatment. We will do this using blood tests and imaging the patients' arteries with ultrasound. We will also measure how cost-effective it is for a hospital to run the program.

It is our goal to develop a community health worker model that is culturally sensitive for people with cultural, educational or educational barriers. Statin use is known to benefit patients in theory; such a culturally competent program will improve health outcomes in practice. After we test it, a cost-effective program such as this can be implemented in other hospitals.

DETAILED DESCRIPTION:
The lipid-specific and pleiotropic benefits of statin therapy, and secondary prevention of coronary artery disease (CAD) mortality have been demonstrated. Statin therapy in particular is underutilized in both white and Black American populations who have CAD and who do not have access to therapy or who cannot afford it. Systems factors related to these findings involve a lack of continuous access to medications following hospital discharge for many Black Americans and for white Americans who do not have the ability to readily afford their medicines or who do not have the educational background to understand the importance of therapy. In many cases, there is failure by primary care physicians to continue statin therapy after discharge in patients who have poor access to therapy or who do not comply with pharmacotherapy. Patient factors include mistrust and volitional nonadherence related to beliefs and personal priorities, and a lack of education and support related to preventive therapy.

This trial will thus take place in lower income and lower educational level Black and white American patients identified at the time of hospitalization and will continue for two years after a myocardial infarction, coronary artery bypass graft, or percutaneous intervention. The overall hypothesis is that a quality of care intervention delivered to Black and white American patients with lower incomes and /or education by a culturally competent community health worker (CHW) within an existing hospital system will result in improved outcomes. The CHW will counsel patients and help them access resources, including Maryland and private pharmacy assistance programs. The specific aims are to compare the impact of a hospital-based CHW intervention versus usual care (UC) on (1) the percent who achieve LDL cholesterol goals, (2) adherence to the statin regimen, and (3) health outcomes including inflammatory markers and vascular function at 6 and 12 months after hospitalization for the premature CAD event. (Participants enrolled during the early phase of the recruitment will have an additional study visit at 24 months.) We will determine the cost of achieving the LDL-C goal in each group. Outcome measures include patient adherence (pill counts, modified Hill-Bone questionnaire), lipid parameters, hs-CRP, and brachial artery reactivity as a marker of endothelial function.

Intention to treat analyses will be used. Multivariable adjusted analysis using generalized linear models or generalized estimating equations will be used to determine the independent effect of the interventions after adjusting for covariates. A sample size of 68 subjects per group can detect hypothesized differences in the proportion of participants meeting goal levels of LDL-C with 92% power, as the primary outcome at 1 years. This proposal will demonstrate the effectiveness of a potentially generalizable model of culturally competent care that will improve the use of statin therapy and its health outcomes in Black and white Americans with documented CAD and poor access to statin pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Johns Hopkins Hospital or Johns Hopkins Bayview Medical Center
* Diagnoses of Myocardial Infarction, unstable angina, percutaneous intervention, coronary artery bypass surgery
* One of the following:

  * Less than a high school education (defined as completion of the 12th grade)
  * No insurance for medications with a household income of $50,000. or less
  * Any difficulty in co-pay even with a household income of >$50,000.

Exclusion Criteria:

* physician contraindicates statin use
* chronic glucocorticosteroid therapy
* autoimmune disease (i.e. lupus erythematosus)
* current chemotherapy or radiation
* immediate life-threatening comorbidity (i.e. HIV-AIDS, end-stage renal disease, or cancer)
* history of hepatic or renal failure
* myositis with creatine kinase (CK) elevations
* any prior adverse response to statin therapy
* statin allergy
* rhabdomyolysis
* pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhananjay Vaidya, MBBS PhD MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial recruited lower income and lower educational level Black and white American patients identified at the time of hospitalization of the Johns Hopkins Medical Institutions for a myocardial infarction, coronary artery bypass graft, or percutaneous intervention.
Pre-assignment Details: Participants were enrolled during their hospitalization. Participants had their randomization visit at 1 month.
Groups:
- Patient Navigator Intervention: Patient Navigator intervention
  Navigation by a health worker : Help provided by health worker to navigate medication access programs
- Information Control: Information control
  Information control : Information about medication access programs provided to the participant and their healthcare provider
Period: Overall Study
Arm/Group | Patient Navigator Intervention | Information Control
Started | 36 | 37
Completed | 27 (For the 6 month endpoint) | 25 (For the 6-month endpoint)
Not Completed | 9 | 12
Not completed — Withdrawal by Subject | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Navigator Intervention | Information Control | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 31 | 58
  >=65 years | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.0) | 55.8 (10.2) | 55.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 20 | 21 | 41
Region of Enrollment [Number; unit: participants]
  United States | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Achievement of LDL-cholesterol Goals
Description: Achieving the goal of an LDL cholesterol level of < 100 mg/dL. For intention to treat analysis the randomization visit status is carried forward if data are missing for the 6-month follow-up visit.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Patient Navigator Intervention | Information Control
Number analyzed (Participants) | 36 | 37
participants | 31 | 29

2. Secondary Outcome: Self-reported Medication Adherence
Description: Only individuals with 6-month follow-up data were included in this analysis
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Patient Navigator Intervention | Information Control
Number analyzed (Participants) | 36 | 37
participants | 16 | 19

ADVERSE EVENTS:
Time Frame: ^ months
Description: 2 individuals were enrolled in the hospital but had adverse events before they had their first study visit: 1 death and 1 myocardial infarction. These individuals were not included in the study.
Arm/Group | Patient Navigator Intervention | Information Control
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 0/36 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No